CLINICAL TRIAL: NCT05615454
Title: Effect of Bio-electromagnetic Energy Regulation Therapy on Erectile Dysfunction in Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Abdulaziz Alzahrani, PhD Candidate, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BEMER
Record Dates: First submitted 2022-11-06; First posted 2022-11-14 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Erectile Dysfunction Due to Diseases Classified Elsewhere; Multiple Sclerosis, Relapsing-Remitting
Keywords: BEMER; Erectile Dysfunction; Multiple Sclerosis; bio-electromagnetic energy regulation therapy
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Erectile Dysfunction; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: The intervention will be provided by a treating therapist who has a clinical experience of more than 13 years. The intervention for both groups will be for three consecutive weeks, five days per week (a total of 15 sessions)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization sequence uses an online https://www.randomizer.org// procedure by an independent person not involved in the study. Matching is done using sequentially numbered, concealed opaque envelopes (SNOSE) for equal distribution of subjects between both therapies (Doig & Simpson, 2005). An independent assessor will assess eligibility by following the inclusion and exclusion criteria for treatment allocation. Then he will collect primary demographic data and conduct all outcome measurements pre-and post-treatment. If the participant is eligible, he chooses a sealed envelope placed in a box and goes to the treating therapist. The treating therapist will be blind to outcome measurements. The participants will be blind to the type of treatment, and the independent assessor will be blind to the participants' group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): (BEMER activated)
  Interventions: Device: bio-electromagnetic energy regulation therapy (BEMER) machine model type: B.BOX CLASSIC, model NO: 420100, 12-15 Volt, (BEMER Int.AG, Liechtenstein product).
- Comparison group (Placebo Comparator): (BEMER deactivated)
  Interventions: Device: placebo BEMER

INTERVENTIONS:
Device: bio-electromagnetic energy regulation therapy (BEMER) machine model type: B.BOX CLASSIC, model NO: 420100, 12-15 Volt, (BEMER Int.AG, Liechtenstein product). — The experimental group (receive the BEMER therapy) for five sessions/week for three weeks. Plus, pelvic floor exercise.
  Arms: Experimental group
Device: placebo BEMER — Comparison group (receive placebo BEMER therapy) for five sessions/week for three weeks. Plus, pelvic floor exercise.
  Arms: Comparison group

SUMMARY:
Multiple sclerosis (MS) is an inflammatory disease that affects the brain and spinal cord. There are potential impacts on neurological functions, including sensory and autonomic functions. The Primary observed in males with MS is erectile dysfunction (ED), which substantially impacts the quality of life. There is increasing literature on electromagnetic fields' biological and clinical effects, particularly on ED.

DETAILED DESCRIPTION:
The study aims to examine the bio-electromagnetic energy regulation therapy (BEMER) on erectile dysfunction with MS. We will recruit participants with MS having ED in a Triple-blind randomized clinical trial study. All participants will be randomly assigned to either an experimental group (receive the BEMER therapy) or a comparison group (receive placebo BEMER therapy) for five days/week for three weeks. Participants will also receive pelvic floor exercises in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS according to the McDonald Revised criteria.
* Score 6-25 on the International Index of Erectile Function 15 (IIEF-15) will be recruited.
* Had sexual activity in the past month.
* Have Relapsing-remitting MS (RRMS) type and one month of clinical relapse, at least before the experimental study date.

Exclusion Criteria:

* If they have cognitive impairment that causes problems in answering the questionnaire.
* History of major chronic illness or other neurological disorders.
* Received any treatment for ED in the past seven days
* Previous therapy with a pulsed electromagnetic field, epilepsy, pacemaker, and acute bacterial infection with fever.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Adult men (18-40 years old)
Enrollment: 50 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
International Index of Erectile Function - Erectile Function (IIEF-EF) | Change from Baseline Erectile Function at 3 weeks
  International Index of Erectile Function Erectile Function domain (IIEF-EF domain score) this means only questions 1, 2, 3, 4, 5, and 15 of IIEF-15.

SECONDARY OUTCOMES:
The Arizona Sexual Experience (ASEX) Scale | Within immediately of completion of the 3-week intervention period.
  The ASEX was designed to assess five significant aspects of sexual dysfunction: drive, arousal, penile erection/vaginal lubrication, capability to achieve orgasm, and orgasmic satisfaction. Items are measured on a 6-point scale (1-6), with higher scores reflecting impaired sexual function. This scale allows for quick detection of sexual dysfunction. Sexual dysfunction was defined as one ASEX total score of ≥19, 2, any one item with a score of 5 or 3, or any three items with a score of ≥4
Modified Fatigue Impact Scale (MFIS) | Within immediately of completion of the 3-week intervention period.
  The MFIS is a 21-item, multidimensional questionnaire that collects information about the effects of physical (9-item), psychosocial (2-item), and cognition (10-item) fatigue over the past four weeks. Participants ranked the 21 items on a 5-point Likert scale with anchors of never (0) and always (4). The optimal cutoff scores of the overall MFIS-A, physical/social, and cognitive subscales indicative of fatigue are 35.5, 18.5, and 15.5, respectively. Changes of 14.68 points or more may indicate a clinically significant change in fatigue in multiple sclerosis patients.
The Multiple Sclerosis, Intimacy, and Sexuality Questionnaire (MSISQ-19) | Within immediately of completion of the 3-week intervention period.
  The MSISQ-19 is the most accurate and widely used tool for exploring the impact of MS on sexual function, assessing all aspects of sexual life and all three levels of sexual dysfunction (Domingo et al., 2018). It is a 19-item self-report questionnaire assessing the effect of MS symptoms on sexual activity and general sexual satisfaction during the previous six months (Carotenuto et al., 2021). Each item is scored on a Likert scale (1=never, 2=rarely, 3=sometimes, 4=often, and 5=always). In addition to the overall score, the MSISQ-19 provides scores on three different subscales: primary sexual dysfunction (calculated by items 12, 16, 17, 18, and 19) , Secondary sexual dysfunction (calculated by items 1, 2, 3, 4, 5, 6, 8, 10, and 11) and tertiary sexual dysfunction (described by items 7, 9, 13, 14, and 15) (Carotenuto et al., 2021)

OTHER OUTCOMES:
Erection Hardness Scale (EHS) | Within immediately of completion of the 3-week intervention period.
  The EHS is used to rate the hardness of a penile erection. The patient will be asked: How would you rate the hardness of your erection? EHS has a 5-point Likert scale from 0 (penis does not enlarge) to 5 (the penis is completely hard and fully rigid)

CONTACTS AND LOCATIONS:
Overall Officials: Abdulaziz A Alzahrani, PhDcandidate, Principal Investigator — imam abdurhman bin faisal
Locations (2):
- Saudi Arabia (2):
  - Ali Muteb Alshami, Dammam
  - Imam Abdulrahman Bin Faisal University, Dammam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdulla FA, Albagmi FM, Al-Khamis FA. Factors that influence quality of life in patients with multiple sclerosis in Saudi Arabia. Disabil Rehabil. 2022 Aug;44(17):4775-4783. doi: 10.1080/09638288.2021.1919929. Epub 2021 May 9. PMID 33966564
- [Background] Alawami AS, Abdulla FA. Psychometric properties of an Arabic translation of the modified fatigue impact scale in patients with multiple sclerosis. Disabil Rehabil. 2021 Nov;43(22):3251-3259. doi: 10.1080/09638288.2020.1731853. Epub 2020 Feb 28. PMID 32109166
- [Background] AlJumah M, Bunyan R, Al Otaibi H, Al Towaijri G, Karim A, Al Malik Y, Kalakatawi M, Alrajeh S, Al Mejally M, Algahtani H, Almubarak A, Cupler E, Alawi S, Qureshi S, Nahrir S, Almalki A, Alhazzani A, Althubaiti I, Alzahrani N, Mohamednour E, Saeedi J, Ishak S, Almudaiheem H, El-Metwally A, Al-Jedai A. Rising prevalence of multiple sclerosis in Saudi Arabia, a descriptive study. BMC Neurol. 2020 Feb 8;20(1):49. doi: 10.1186/s12883-020-1629-3. PMID 32035478
- [Background] Ben-Zacharia AB. Therapeutics for multiple sclerosis symptoms. Mt Sinai J Med. 2011 Mar-Apr;78(2):176-91. doi: 10.1002/msj.20245. PMID 21425263
- [Background] Carotenuto A, De Giglio L, Chiodi A, Petracca M, Rosa L, Bianchi M, Ferrante I, Lauro F, Moccia M, Ianniello A, Pozzilli C, Brescia Morra V, Lanzillo R. Validation of the Italian version of the Multiple Sclerosis Intimacy and Sexuality Questionnaire-19. Neurol Sci. 2021 Jul;42(7):2903-2910. doi: 10.1007/s10072-020-04873-w. Epub 2020 Nov 21. PMID 33222102
- [Background] Compston A, Coles A. Multiple sclerosis. Lancet. 2008 Oct 25;372(9648):1502-17. doi: 10.1016/S0140-6736(08)61620-7. PMID 18970977
- [Background] Dastoorpoor M, Zamanian M, Moradzadeh R, Nabavi SM, Kousari R. Prevalence of sexual dysfunction in men with multiple sclerosis: a systematic review and meta-analysis. Syst Rev. 2021 Jan 6;10(1):10. doi: 10.1186/s13643-020-01560-x. PMID 33407874
- [Background] Doig GS, Simpson F. Randomization and allocation concealment: a practical guide for researchers. J Crit Care. 2005 Jun;20(2):187-91; discussion 191-3. doi: 10.1016/j.jcrc.2005.04.005. PMID 16139163
- [Background] Dorey G, Speakman M, Feneley R, Swinkels A, Dunn C, Ewings P. Randomised controlled trial of pelvic floor muscle exercises and manometric biofeedback for erectile dysfunction. Br J Gen Pract. 2004 Nov;54(508):819-25. PMID 15527607
- [Background] Dorey G, Speakman MJ, Feneley RC, Swinkels A, Dunn CD. Pelvic floor exercises for erectile dysfunction. BJU Int. 2005 Sep;96(4):595-7. doi: 10.1111/j.1464-410X.2005.05690.x. PMID 16104916
- [Background] Gandhi F, Jhaveri S, Avanthika C, Singh A, Jain N, Gulraiz A, Shah P, Nasir F. Impact of Vitamin D Supplementation on Multiple Sclerosis. Cureus. 2021 Oct 5;13(10):e18487. doi: 10.7759/cureus.18487. eCollection 2021 Oct. PMID 34754649
- [Background] Gerbild H, Larsen CM, Graugaard C, Areskoug Josefsson K. Physical Activity to Improve Erectile Function: A Systematic Review of Intervention Studies. Sex Med. 2018 Jun;6(2):75-89. doi: 10.1016/j.esxm.2018.02.001. Epub 2018 Apr 13. PMID 29661646
- [Background] Goldstein I, Lue TF, Padma-Nathan H, Rosen RC, Steers WD, Wicker PA. Oral sildenafil in the treatment of erectile dysfunction. Sildenafil Study Group. N Engl J Med. 1998 May 14;338(20):1397-404. doi: 10.1056/NEJM199805143382001. PMID 9580646
- [Background] Gyulai F, Raba K, Baranyai I, Berkes E, Bender T. BEMER Therapy Combined with Physiotherapy in Patients with Musculoskeletal Diseases: A Randomised, Controlled Double Blind Follow-Up Pilot Study. Evid Based Complement Alternat Med. 2015;2015:245742. doi: 10.1155/2015/245742. Epub 2015 May 20. PMID 26078768
- [Background] Kalyvianakis D, Hatzichristou D. Low-Intensity Shockwave Therapy Improves Hemodynamic Parameters in Patients With Vasculogenic Erectile Dysfunction: A Triplex Ultrasonography-Based Sham-Controlled Trial. J Sex Med. 2017 Jul;14(7):891-897. doi: 10.1016/j.jsxm.2017.05.012. PMID 28673433
- [Background] Kanaparthi A, Kesary SPR, Pujita C, Gopalaiah H. Bio Electro Magnetic Energy Regulation (BEMER) therapy in myofascial pain dysfunction syndrome: A preliminary study. J Oral Biol Craniofac Res. 2020 Apr-Jun;10(2):38-42. doi: 10.1016/j.jobcr.2020.01.007. Epub 2020 Feb 3. PMID 32090003
- [Background] Keller JJ, Liang YC, Lin HC. Association between multiple sclerosis and erectile dysfunction: a nationwide case-control study. J Sex Med. 2012 Jul;9(7):1753-9. doi: 10.1111/j.1743-6109.2012.02746.x. Epub 2012 Apr 30. PMID 22548978
- [Background] Lappin MS, Lawrie FW, Richards TL, Kramer ED. Effects of a pulsed electromagnetic therapy on multiple sclerosis fatigue and quality of life: a double-blind, placebo controlled trial. Altern Ther Health Med. 2003 Jul-Aug;9(4):38-48. PMID 12868251
- [Background] Li V, Haslam C, Pakzad M, Brownlee WJ, Panicker JN. A practical approach to assessing and managing sexual dysfunction in multiple sclerosis. Pract Neurol. 2020 Apr;20(2):122-131. doi: 10.1136/practneurol-2019-002321. Epub 2019 Nov 21. PMID 31753860
- [Background] Marck CH, Jelinek PL, Weiland TJ, Hocking JS, De Livera AM, Taylor KL, Neate SL, Pereira NG, Jelinek GA. Sexual function in multiple sclerosis and associations with demographic, disease and lifestyle characteristics: an international cross-sectional study. BMC Neurol. 2016 Nov 4;16(1):210. doi: 10.1186/s12883-016-0735-8. PMID 27814701
- [Background] Moussa M, Abou Chakra M, Papatsoris AG, Dabboucy B, Hsieh M, Dellis A, Fares Y. Perspectives on urological care in multiple sclerosis patients. Intractable Rare Dis Res. 2021 May;10(2):62-74. doi: 10.5582/irdr.2021.01029. PMID 33996350
- [Background] Nakhli J, El Kissi Y, Bouhlel S, Amamou B, Nabli TA, Nasr SB, Ali BB. Reliability and validity of the Arizona sexual experiences scale-Arabic version in Tunisian patients with schizophrenia. Compr Psychiatry. 2014 Aug;55(6):1473-7. doi: 10.1016/j.comppsych.2014.04.006. Epub 2014 Apr 12. PMID 24850067
- [Background] Palm P, Zwisler AO, Svendsen JH, Thygesen LC, Giraldi A, Jensen KG, Lindschou J, Winkel P, Gluud C, Steinke E, Berg SK. Sexual rehabilitation for cardiac patients with erectile dysfunction: a randomised clinical trial. Heart. 2019 May;105(10):775-782. doi: 10.1136/heartjnl-2018-313778. Epub 2018 Oct 31. PMID 30381319
- [Background] Pelka RB, Jaenicke C, Gruenwald J. Impulse magnetic-field therapy for erectile dysfunction: a double-blind, placebo-controlled study. Adv Ther. 2002 Jan-Feb;19(1):53-60. doi: 10.1007/BF02850018. PMID 12008861
- [Background] Polman CH, Reingold SC, Edan G, Filippi M, Hartung HP, Kappos L, Lublin FD, Metz LM, McFarland HF, O'Connor PW, Sandberg-Wollheim M, Thompson AJ, Weinshenker BG, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2005 revisions to the "McDonald Criteria". Ann Neurol. 2005 Dec;58(6):840-6. doi: 10.1002/ana.20703. PMID 16283615
- [Background] Rennie D. CONSORT revised--improving the reporting of randomized trials. JAMA. 2001 Apr 18;285(15):2006-7. doi: 10.1001/jama.285.15.2006. No abstract available. PMID 11308440
- [Background] Rosen RC, Cappelleri JC, Gendrano N 3rd. The International Index of Erectile Function (IIEF): a state-of-the-science review. Int J Impot Res. 2002 Aug;14(4):226-44. doi: 10.1038/sj.ijir.3900857. PMID 12152111
- [Background] Rosenbaum TY. Pelvic floor involvement in male and female sexual dysfunction and the role of pelvic floor rehabilitation in treatment: a literature review. J Sex Med. 2007 Jan;4(1):4-13. doi: 10.1111/j.1743-6109.2006.00393.x. PMID 17233772
- [Background] Shafik A, el-Sibai O, Shafik AA. Magnetic stimulation of the cavernous nerve for the treatment of erectile dysfunction in humans. Int J Impot Res. 2000 Jun;12(3):137-41; discussion 141-2. doi: 10.1038/sj.ijir.3900521. PMID 11045905
- [Background] Shamloul R, Ghanem H, Abou-zeid A. Validity of the Arabic version of the sexual health inventory for men among Egyptians. Int J Impot Res. 2004 Oct;16(5):452-5. doi: 10.1038/sj.ijir.3901248. PMID 15175638
- [Background] Thomas C, Konstantinidis C. Neurogenic Erectile Dysfunction. Where Do We Stand? Medicines (Basel). 2021 Jan 7;8(1):3. doi: 10.3390/medicines8010003. PMID 33430218
- [Background] Vardi Y, Appel B, Jacob G, Massarwi O, Gruenwald I. Can low-intensity extracorporeal shockwave therapy improve erectile function? A 6-month follow-up pilot study in patients with organic erectile dysfunction. Eur Urol. 2010 Aug;58(2):243-8. doi: 10.1016/j.eururo.2010.04.004. Epub 2010 May 6. PMID 20451317